CLINICAL TRIAL: NCT04308954
Title: Cross-Species Multi-Modal Neuroimaging to Investigate GABA Physiology in Fragile X Syndrome
Brief Title: Neuroimaging GABA Physiology in Fragile X Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty with patient recruitment due to COVID-19 pandemic
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Frederick Chin, PhD, Assistant Professor (Research) of Radiology (General Radiology), Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB 32149
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Fragile X Syndrome (FXS); Idiopathic Intellectual Developmental Disorder (IDD)
Keywords: FXS, Intellectual Disability
MeSH Terms: conditions — Fragile X Syndrome; Intellectual Disability | interventions — 5-(2'-fluoroethyl)flumazenil

STUDY DESIGN:
Intervention Model Description: 15 male subjects with FXS will be compared to 15 subjects with idiopathic intellectual developmental disorder, who will be the control group. Young male adults with idiopathic intellectual developmental disorder will be (group) matched to FXS participants for mean age (and age range), handedness, socioeconomic status and ethnicity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fragile X Syndrome (Experimental): Adult males aged 18-30 years diagnosed with FXS will undergo a non-invasive F18 FMZ PET/MRI scan to determine GABA(A) receptor density; developmental dynamics of GABA(A) receptor distribution, and structural neuroanatomy and connectional anatomy.
  Interventions: Drug: [18F]flumazenil
- Idiopathic Intellectual Developmental Disorder (Experimental): Adult males aged 18-30 years diagnosed with idiopathic intellectual developmental disorder will undergo a non-invasive F18 FMZ PET/MRI scan to determine GABA(A) receptor density; developmental dynamics of GABA(A) receptor distribution, and structural neuroanatomy and connectional anatomy.
  Interventions: Drug: [18F]flumazenil

INTERVENTIONS:
Drug: [18F]flumazenil — [18F]flumazenil is a PET radiopharmaceutical that can be used to determine gamma-aminobutyric acid (GABA(A)) receptor density.
  Other Names: F18 FMZ

SUMMARY:
The investigators wish to compare the brain distribution of GABA(A) receptors and GABA levels in young adult males with Fragile X Syndrome compared to idiopathic intellectual developmental disorder. The radiopharmaceutical [18F]flumazenil has been used to study GABA(A) receptor distribution in other genetic syndromes with autistic features; however, despite overwhelming evidence supporting the importance of the GABAergic system in FXS, no clinical investigation of this system in human FXS has been reported in the literature. Therefore, this study will provide the first in vivo comprehensive examination of the GABAergic system in FXS using hybrid positron emission tomography/ magnetic resonance imaging (PET/MRI).

DETAILED DESCRIPTION:
Fragile X syndrome (FXS) is the most common genetic cause of autism spectrum disorder (ASD). Converging evidence suggests that GABAergic dysfunction occurs in FXS. The investigators wish to examine brain distribution of GABA (A) receptors in young adult males with FXS using hybrid PET/MRI with [18F]flumazenil. This project will study the distribution of GABA(A) receptors in 15 young male adults with FXS (18-30 years old) compared to 15 age-matched male subjects with idiopathic intellectual developmental disorder (IDD) as controls. Simultaneous PET/MRI acquisition is an optimal technique to study in vivo GABAergic dysfunction and GABAa receptor distribution.

ELIGIBILITY:
Inclusion Criteria for participants with FXS:

1. Have an established diagnosis of FXS (full mutation with aberrant FMR1 methylation) by genetic testing
2. Diagnosis of intellectual disability
3. Males who are physically healthy
4. Age 18 to 30 years inclusive
5. IQ between 40 and 80 points
6. Ability to remain seated for more than 10 minutes
7. Ability to travel to Stanford

Exclusion criteria for participants with FXS:

1. Diagnosis of a known genetic disorder (other than FXS).
2. Active medical problems such as unstable seizures, congenital heart disease, endocrine disorders.
3. Significant sensory impairments such as blindness or deafness.
4. DSM-5 diagnosis of other severe psychiatric disorder such as bipolar disorder or schizophrenia.
5. Pre-term birth (<34 weeks' gestation) or low birth weight (<2000g).
6. Current use of benzodiazepines.
7. Contraindication for PET or MRI.

Inclusion criteria for participants with IDD:

1. Age 18 to 30 years inclusive
2. Adults who are physically healthy
3. No significant recent changes in psychosocial stressors per history
4. Diagnosis of intellectual disability
5. IQ between 40 and 80 points
6. Ability to remain seated for more than 10 minutes
7. Ability to travel to Stanford

Exclusion Criteria for participants with IDD:

1. Genetic diagnosis of FXS.
2. Active medical problems such as unstable seizures, congenital heart disease, endocrine disorders.
3. Significant sensory impairments such as blindness or deafness.
4. DSM-5 diagnosis of other severe psychiatric disorder such as bipolar disorder or schizophrenia.
5. Pre-term birth (<34 weeks' gestation) or low birth weight (<2000g).
6. Current use of benzodiazepines.
7. Contraindication for PET or MRI.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participants must be male adults with idiopathic intellectual developmental disorder (IDD) or fragile X-syndrome (FXS)
Enrollment: 17 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Non-displaceable binding potential of [18F]flumazenil (F18 FMZ) | Up to 2 hours per scan on a single study day
  Binding potential provides an estimate of the GABA (A) receptor distribution and affinity of [18F]flumazenil-PET to the GABA receptors. Binding potential will be measured in patients with fragile X syndrome and control group comprising individuals with idiopathic intellectual developmental disorder.
  Using imaging data obtained from PET that was corrected for attenuation and partial volume effects by MRI, nuclear medicine physicians will draw regions of interest (ROI's) around the areas of the brain listed below to estimate the F18 FMZ non-displaceable binding potential (BPnd) of F18 FMZ to GABA (A) receptors in FXS.
GABA (A) receptor density in fragile X syndrome (FXS) patients relative to control group comprising individuals with idiopathic Intellectual Developmental Disorder (IDD) | Up to 2 hours per scan on a single study day
  Binding potential measurements will be compared between participants with fragile X syndrome and control group with idiopathic intellectual developmental disorder(IDD) using the PET radiotracer [18F]flumazenil-PET.
  Binding Potential (BPnd) is estimated as the distribution volume ratio (DVR) -1.
  DVR's of tracers are used in PET receptor studies where the radiopharmaceutical can be specifically bound to receptors; nonspecifically bound to other macromolecular components, or free in tissue (FT). DVR is calculated using a Logan Plot, which uses the dynamic PET images obtained during imaging and compartment modeling to graphically analyze by linear regression pharmacokinetic data for radiopharmaceuticals that undergo 'reversible' uptake.
  PET scans of FXS patients will be compared to the PET scans of control group.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick T Chin, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lucignani G, Panzacchi A, Bosio L, Moresco RM, Ravasi L, Coppa I, Chiumello G, Frey K, Koeppe R, Fazio F. GABA A receptor abnormalities in Prader-Willi syndrome assessed with positron emission tomography and [11C]flumazenil. Neuroimage. 2004 May;22(1):22-8. doi: 10.1016/j.neuroimage.2003.10.050. PMID 15109994
- [Background] Holopainen IE, Metsahonkala EL, Kokkonen H, Parkkola RK, Manner TE, Nagren K, Korpi ER. Decreased binding of [11C]flumazenil in Angelman syndrome patients with GABA(A) receptor beta3 subunit deletions. Ann Neurol. 2001 Jan;49(1):110-3. doi: 10.1002/1531-8249(200101)49:13.0.co;2-t. PMID 11198279